CLINICAL TRIAL: NCT04669678
Title: An Observational Pharmacokinetic Study to Evaluate Drug-drug Interactions Between Doravirine-containing ART and Hormonal Contraceptives Among Women Living With HIV in South Africa.
Brief Title: Evaluation of Pharmacokinetic Drug-drug Interactions Between Hormonal Contraceptives and Doravirine-containing ART Among Women Living With HIV in South Africa
Acronym: EPIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Wits Reproductive Health and HIV Institute (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Rena Patel, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00011487; MISP 59559 (Other Grant/Funding Number: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2020-11-25; First posted 2020-12-17 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections; Contraception; Drug-drug Interaction
MeSH Terms: conditions — HIV Infections | interventions — etonogestrel

STUDY DESIGN:
Intervention Model Description: Different groups receive different interventions at same time during study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group 1 DOR + ETG (Experimental): 100mg DOR-containing ART [oral tablet taken daily] + 68mg ETG implant (follow up for 30 weeks)
  Interventions: Drug: Etonogestrel (ETG) implant
- Group 2 DOR + IM DMPA (Experimental): 100mg DOR-containing ART [oral tablet taken daily] + 150mg IM DMPA (follow up for 18 weeks)
  Interventions: Drug: Intramuscular depo-medroxyprogesterone acetate (IM DMPA)
- Group 3 DOR + SC MPA (Experimental): 100mg DOR-containing ART [oral tablet taken daily] + 104mg SC MPA (follow up for 18 weeks)
  Interventions: Drug: Sub-cutaneous medroxyprogesterone acetate (SC MPA)
- Group 4 DOR + IUD (Experimental): 100mg DOR-containing ART [oral tablet taken daily] + 1 non-hormonal IUD device (follow up for 30 weeks)
  Interventions: Device: Non-hormonal intrauterine device (IUD)
- Group 5 DTG + DMPA (Active Comparator): 50mg DTG-containing ART [oral tablet taken daily] + 150mg IM DMPA DMPA administered at enrolment (follow up for 18 weeks)
  Interventions: Drug: Intramuscular depo-medroxyprogesterone acetate (IM DMPA)

INTERVENTIONS:
Drug: Etonogestrel (ETG) implant — Contraceptive progestin implants are thin rods inserted under the skin of a woman's arm. The most widely available implant in South Africa is currently Implanon®/Nexplanon®/Implanon NXT®, containing etonogestrel (ETG, 3-keto desogestrel). Implanon® consists of a single rod of ethylene vinyl acetate and contains 68 mg of ETG; it is manufactured by Merck and is approved for 3 years.
  Arms: Group 1 DOR + ETG
Drug: Intramuscular depo-medroxyprogesterone acetate (IM DMPA) — DMPA (150 mg of depo-medroxyprogesterone acetate (MPA)/ml IMI) is the most commonly used injectable contraceptive worldwide, and the most commonly used method of reversible injectable contraception in sub-Saharan Africa.
  Arms: Group 2 DOR + IM DMPA; Group 5 DTG + DMPA
Drug: Sub-cutaneous medroxyprogesterone acetate (SC MPA) — SC MPA or Sayana® Press is a single-dose container with 104 mg medroxyprogesterone acetate (MPA) in 0.65 mL suspension for injection. Sayana® Press is indicated for medium-long term female contraception.
  Arms: Group 3 DOR + SC MPA
Device: Non-hormonal intrauterine device (IUD) — The NOVA T-380 non-hormonal IUD consists of a T-shaped polyethylene frame wound with copper wire, along with two monofilament threads to aid in removal of the IUD. IUDs may be left in place for up to 5 years.
  Arms: Group 4 DOR + IUD

SUMMARY:
The study investigators are conducting an observational, parallel group pharmacokinetic (PK) study among women living with HIV (WLHIV) already on 1st line antiretroviral therapy (ART) and virally suppressed, 18-45 years old (inclusive), to evaluate any bidirectional drug-drug interactions (DDIs) between doravirine (DOR)-containing ART and hormonal contraceptive methods. This PK study will enroll women in five distinct groups, each with 21 participants (total of 105 participants), and follow them for approximately 18-30 weeks.

DETAILED DESCRIPTION:
While DOR-containing ART has been evaluated in two large clinical trials, only 16-17% of the study participants were women and only 6-10% of them were African. In an epidemic, where the gendered majority affected by the disease are women of reproductive age living in Africa, it is imperative to conduct a study evaluating reproductive health outcomes among and specific to African women. Further underscoring the issue is a notable data gap for DOR regarding DDIs with the most common leading hormonal contraceptives.

Our intention is to study potential DDIs between DOR and the most common contraceptive methods used by WLHIV in an African context, which generally include short- (e.g., OCPs/COCs), intermediate (e.g., injectable) or long-acting (e.g., implants or IUDs) methods. Since the drug maker of DOR has already conducted the industry standard PK study with DOR and a COC product, containing ethinyl estradiol and levonorgestrel, which did not demonstrate any bidirectional DDI, the investigators have chosen to exclude this method from the current study. Thus, the current EPIC study focuses on intermediate- and long-acting contraceptive methods, which have different PK profiles than daily administrated oral drugs and may be more susceptible to potential DDIs with DOR.

Participants who are interested in self-selecting and initiating one of the study contraceptive methods listed will be recruited for screening and eligibility assessments. If eligible and enrolled, there will be a 6-week lead-in period with daily use of oral DOR-containing ART followed by contraceptive method initiation of their choice. Study follow-up will take place every 2-4 weeks, at a minimum, for an additional 12 or 24 weeks for a total of 18 or 30 weeks of follow-up depending on the contraceptive method chosen.

The investigators will also enroll a dolutegravir (DTG) + IM DMPA group, who will be followed for 12 weeks, as the comparator group for the DOR + IM DMPA group.

The comparator group for the DOR + etonogestrel (ETG) implant group will be a historical control group from a similar PK study called PARVI (PK study of ARVs and Implants in Kenya) that is currently being conducted by Dr. Patel and colleagues in Kenya.

The five study groups are summarized below in Table 1.

Table 1: Study groups by ART regimen and contraceptive method choice

Group number N ART regimen and contraceptive method Group 1 21 DOR-containing ART + initiating ETG implant Group 2 21 DOR-containing ART + initiating IM DMPA Group 3 21 DOR-containing ART + initiating SC MPA Group 4 21 DOR-containing ART + initiating non-hormonal IUD Group 5 21 DTG-containing ART + initiating IM DMPA

The co-primary objectives are to evaluate any associations between doravirine (DOR), a newer antiretroviral agent for the treatment of HIV, exposure and hormonal contraceptive use in the four groups of DOR + 1) etonogestrel implant (ETG), 2) intramuscular depomedroxyprogesterone acetate (IM DMPA), 3) subcutaneous medroxyprogesterone acetate (SC MPA), or 4) non-hormonal IUD users by generating mean hormone concentrations at 12 weeks for IM and SC DMPA or 24 weeks for ETG implants and IUD groups; also to evaluate any bi-directional associations between hormonal contraceptive exposure and DOR use by generating mean DOR concentration at 24 hours.

The first hypotheses are: the mean implant hormone concentrations for DOR + ETG implant at 24 weeks after implant placement will be similar (i.e. geometric mean ratio [GMR] within 0.80 and 1.25) to the mean implant hormone concentrations for DTG + ETG implant (historical controls from Dr. Patel's current PARVI study in a similar population in Kenya). The mean MPA concentrations for DOR + IM DMPA or SC MPA at 12 weeks after DMPA/MPA administration will be similar (i.e. GMR within 0.8 and 1.25) to the mean DMPA concentrations for DTG + DMPA (contemporaneous study group). Also, the mean C24 hours of DOR in the ETG implant and MPA groups will be similar to the non-hormonal contraceptive method (i.e. the non-hormonal IUD) group.

The secondary objectives are to measure DOR-containing ART's efficacy, via HIV viral load <40 copies/mL, at 12-24 weeks after contraceptive initiation among women of reproductive age using hormonal and non-hormonal contraceptives.

The second hypothesis is that proportion of women suppressed (defined as HIV viral load <40 copies/mL) at 16-30 weeks after DOR-containing ART initiation will be similar to a contemporaneous or historical comparison of the proportion of women suppressed with non-DOR containing ART from the same study population/sample.

The exploratory objectives are to qualitatively explore decision-making around ART and contraceptive options, study experiences of ART switch, and use of the contraceptive method, including self-administration of SC MPA, and to describe self-reported experiences of social harms and social benefits related to study participation. Also, safety including side effects, satisfaction, and continuation rates of both the hormonal contraceptive method and ART will be assessed.

The third hypothesis is that the safety, satisfaction, and continuation rates of the various contraceptive methods will be similar to each other at 12-24 weeks after contraceptive initiation. The investigators will gain interesting insights into women's decision-making around ART and contraceptive method options and are uniquely positioned to describe experiences of self-administration of SC MPA.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Currently on 1st line ART (namely EFV- or DTG-containing ART),
* Have documented or confirmed viral suppression for HIV (defined as <40 copies/mL) within 3 months prior to study screening and after the start of the current ART regimen
* Contraception use:

  a) Not currently on reliable contraception and intending to or willing to initiate use of study hormonal/non-hormonal contraceptive methods 6 weeks after DOR lead in period (and willing to continue use for subsequent 12 to 24 weeks),
* Able and willing to comply with all study procedural requirements,
* Able and willing to provide informed consent for study participation in either English or Zulu,
* Able and willing to provide adequate locator information, as defined in site SOPs,
* Negative pregnancy test at Screening and Enrollment, and
* At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, or vaccines for the duration of study participation.

Exclusion Criteria:

* Currently on 2nd line, 3rd line, or salvage ART regimens,
* Currently pregnant or intending to become pregnant within the next 6 months,
* Currently breastfeeding or intending to breastfeed within the next 6 months,
* Use or anticipated use of drugs for the duration of the study period known to interact with hormonal implants, DMPA/MPA, or the respective ART regimen
* Current or planned concomitant use of other hormonal contraceptives,
* Currently obese (BMI≥30),
* Has any of the following laboratory abnormalities at Screening Visit:

  1. Haemoglobin abnormality Grade 2 or higher
  2. Calculated creatinine clearance less than 50 mL/min by the Schwartz Equation
* Per participant report at Screening and Enrollment, intends to do any of the following during her study participation period:

  1. relocate away from the study site
  2. travel away from the study site for a time period that would interfere with product resupply and study participation
* Per participant report and/or clinical evidence of any of the following:

  1. Known adverse reaction to any of the study products (ever),
  2. Participation in any other research study involving drugs, medical devices or vaccines within 60 days of enrollment,
  3. At Enrollment, as determined by the PI/designee, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder, metabolic bone disease or infectious disease,
* We will test for hepatitis B and if participant has the infection, they will be excluded from the study. We also will test for hepatitis B immunity and the participant is not immune, we will offer the vaccination against hepatitis B infection.
* Has any other condition that, in the opinion of the PI/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, MPH, Study Chair — University of Washington; Thesla Palanee-Phillips, MMed Sci PhD, Principal Investigator — Wits Reproductive Health and HIV Institute, Research Centre Clinical Research Site
Locations (1):
- Wits Reproductive Health and HIV Institute, Research Centre Clinical Research Site, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patel RC, Stalter R, Onono M, et al. Dolutegravir-containing ART does not reduce etonogestrel implant concentrations. Conference on Retroviruses and Opportunistic Infections (CROI); March 8-11, 2020; Virtual (Boston).
- [Background] Orkin C, Squires KE, Molina JM, Sax PE, Wong WW, Sussmann O, Kaplan R, Lupinacci L, Rodgers A, Xu X, Lin G, Kumar S, Sklar P, Nguyen BY, Hanna GJ, Hwang C, Martin EA; DRIVE-AHEAD Study Group. Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate is Non-inferior to Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate in Treatment-naive Adults With Human Immunodeficiency Virus-1 Infection: Week 48 Results of the DRIVE-AHEAD Trial. Clin Infect Dis. 2019 Feb 1;68(4):535-544. doi: 10.1093/cid/ciy540. PMID 30184165
- [Background] Molina JM, Squires K, Sax PE, Cahn P, Lombaard J, DeJesus E, Lai MT, Xu X, Rodgers A, Lupinacci L, Kumar S, Sklar P, Nguyen BY, Hanna GJ, Hwang C; DRIVE-FORWARD Study Group. Doravirine versus ritonavir-boosted darunavir in antiretroviral-naive adults with HIV-1 (DRIVE-FORWARD): 48-week results of a randomised, double-blind, phase 3, non-inferiority trial. Lancet HIV. 2018 May;5(5):e211-e220. doi: 10.1016/S2352-3018(18)30021-3. Epub 2018 Mar 25. PMID 29592840

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 DOR + ETG | Group 2 DOR + IM DMPA | Group 3 DOR + SC MPA | Group 4 DOR + IUD | Group 5 DTG + DMPA
Started | 23 | 21 | 24 | 21 | 21
Completed | 21 | 21 | 22 | 19 | 21
Not Completed | 2 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 DOR + ENG Implant: 100mg DOR-containing ART [oral tablet taken daily] + 68mg ETG implant (follow up for 30 weeks)
  Etonogestrel (ENG) implant: Contraceptive progestin implants are thin rods inserted under the skin of a woman's arm. The most widely available implant in South Africa is currently Implanon®/Nexplanon®/Implanon NXT®, containing etonogestrel (ENG, 3-keto desogestrel). Implanon® consists of a single rod of ethylene vinyl acetate and contains 68 mg of ENG; it is manufactured by Merck and is approved for 3 years.
- Total: Total of all reporting groups
Arm/Group | Group 1 DOR + ENG Implant | Group 2 DOR + IM DMPA | Group 3 DOR + SC MPA | Group 4 DOR + IUD | Group 5 DTG + DMPA | Total
Number analyzed (Participants) | 21 | 21 | 22 | 19 | 21 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 22 | 19 | 21 | 104
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [28 to 40] | 35 [28 to 38] | 37 [28.2 to 40] | 37 [31 to 42] | 39 [35 to 41] | 37 [29 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 22 | 19 | 21 | 104
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black race | 21 | 21 | 22 | 19 | 21 | 104
Region of Enrollment [Number; unit: participants]
  South Africa | 21 | 21 | 22 | 19 | 21 | 104

OUTCOME MEASURES:

1. Primary Outcome: Hormonal Contraceptive Concentrations
Description: Mean hormone concentrations
Time Frame: at 2,4,8,12 weeks for IM DMPA and SC MPA or 2,4,8,12,20,24 weeks for ETG implants and IUD groups after contraceptive method initiation
Population: Data was collected at 2,4,8,12, 20 and 24 weeks for Group 1 DOR + ETG; at 2,4,8, and 12 weeks for Group 2 DOR + IM DMPA; at 2,4,8, and 12 weeks for Group 3 DOR SC MPA ; at 2,4,8 and 12 weeks for Group 5 DTG+DMPA. The Group 4 DOR+IUD group was not analyzed for hormonal concentrations as the group involves non-hormonal contraception, as per planned statistical analyses.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Group 1 DOR + ETG | Group 2 DOR + IM DMPA | Group 3 DOR + SC MPA | Group 4 DOR + IUD | Group 5 DTG + DMPA
Number analyzed (Participants) | 21 | 21 | 22 | 0 | 21
pg/mL
  Week 2: number analyzed (Participants) | 17 | 20 | 21 | 0 | 20
  Week 2 | 589 [193 to 954] | 1293 [2 to 2852] | 542 [198 to 1067] |  | 1761 [577 to 3610]
  Week 4 | 550 [157 to 4014] | 1047 [514 to 3913] | 412 [156 to 1091] |  | 1283 [384 to 4098]
  Week 8: number analyzed (Participants) | 20 | 20 | 22 | 0 | 21
  Week 8 | 519 [163 to 2827] | 805 [222 to 2310] | 321 [101 to 658] |  | 984 [148 to 2136]
  Week 12: number analyzed (Participants) | 19 | 21 | 19 | 0 | 20
  Week 12 | 475 [85 to 953] | 535 [295 to 1439] | 271 [116 to 523] |  | 602 [13 to 3569]
  Week 20: number analyzed (Participants) | 19 | 0 | 0 | 0 | 0
  Week 20 | 390 [196 to 819] |  |  |  |
  Week 24: number analyzed (Participants) | 21 | 0 | 0 | 0 | 0
  Week 24 | 378 [111 to 521] |  |  |  |
Statistical Analysis 1: Comparison: Group 2 DOR + IM DMPA vs Group 5 DTG + DMPA; Week 2; Test type: Other; p = 0.306, Mixed Models Analysis; Odds Ratio (OR) = 0.85, 90% CI 2-sided [0.65 to 1.11]
Statistical Analysis 2: Comparison: Group 2 DOR + IM DMPA vs Group 5 DTG + DMPA; Week 4; Test type: Other; p = 0.874, Mixed Models Analysis; Odds Ratio (OR) = 0.81, 90% CI 2-sided [0.60 to 1.09]
Statistical Analysis 3: Comparison: Group 2 DOR + IM DMPA vs Group 5 DTG + DMPA; Week 8; Test type: Other; p = 0.646, Mixed Models Analysis; Odds Ratio (OR) = 1.04, 90% CI 2-sided [0.91 to 1.19]
Statistical Analysis 4: Comparison: Group 2 DOR + IM DMPA vs Group 5 DTG + DMPA; Week 12; Test type: Other; p = 0.869, Mixed Models Analysis; Odds Ratio (OR) = 1.02, 90% CI 2-sided [0.82 to 1.28]
Statistical Analysis 5: Comparison: Group 2 DOR + IM DMPA vs Group 3 DOR + SC MPA; Week 2; Test type: Other; p = 0.044, Mixed Models Analysis; Odds Ratio (OR) = 0.51, 90% CI 2-sided [0.30 to 0.88]
Statistical Analysis 6: Comparison: Group 2 DOR + IM DMPA vs Group 3 DOR + SC MPA; Week 4; Test type: Other; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 0.36, 90% CI 2-sided [0.28 to 0.46]
Statistical Analysis 7: Comparison: Group 2 DOR + IM DMPA vs Group 3 DOR + SC MPA; Week 8; Test type: Other; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 0.37, 90% CI 2-sided [0.27 to 0.49]
Statistical Analysis 8: Comparison: Group 2 DOR + IM DMPA vs Group 3 DOR + SC MPA; Week 12; Test type: Other; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 0.44, 90% CI 2-sided [0.35 to 0.54]

2. Primary Outcome: DOR Concentrations
Description: Mean DOR concentration at 24 hours (C24 hours)
Time Frame: at 2,4,8,12 weeks for IM and SC DMPA or 2,4,8,12,20,24 weeks for ETG implants and IUD groups after contraceptive method initiation
Population: Data was collected at 2,4,8,12, 20 and 24 weeks for Group 1 DOR + ETG; at 2,4,8, and 12 weeks for Group 2 DOR + IM DMPA; at 2,4,8, and 12 weeks for Group 3 DOR + SC MPA ; at 2,4,8 and 12 weeks for Group 4 DOR + IUD. The Group 5 DTG + DMPA group was not analyzed for doravirine(DOR) concentrations as the group involves DTG instead of DOR, as per planned statistical analyses.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Group 1 DOR + ETG | Group 2 DOR + IM DMPA | Group 3 DOR + SC MPA | Group 4 DOR + IUD | Group 5 DTG + DMPA
Number analyzed (Participants) | 21 | 21 | 22 | 19 | 0
ng/mL
  Week 2: number analyzed (Participants) | 14 | 16 | 18 | 13 | 0
  Week 2 | 706 [26 to 2852] | 609 [30 to 1752] | 836 [62 to 1653] | 414 [24 to 1472] |
  Week 4: number analyzed (Participants) | 20 | 15 | 18 | 12 | 0
  Week 4 | 897 [268 to 1773] | 906 [101 to 1500] | 770 [368 to 2142] | 785 [34 to 1381] |
  Week 8: number analyzed (Participants) | 15 | 15 | 17 | 9 | 0
  Week 8 | 916 [36 to 2769] | 778 [213 to 1167] | 1002 [58 to 1833] | 894 [61 to 1168] |
  Week 12: number analyzed (Participants) | 17 | 11 | 15 | 12 | 0
  Week 12 | 976 [546 to 2853] | 1068 [476 to 1513] | 1141 [509 to 2712] | 650 [49 to 984] |
  Week 20: number analyzed (Participants) | 11 | 0 | 0 | 13 | 0
  Week 20 | 919 [83.5 to 1522] |  |  | 948 [183 to 1756] |
  Week 24: number analyzed (Participants) | 13 | 0 | 0 | 14 | 0
  Week 24 | 1147 [188 to 1916] |  |  | 766 [262 to 1006] |
Statistical Analysis 1: Comparison: Group 2 DOR + IM DMPA vs Group 4 DOR + IUD; Week 2; Test type: Other; p = 0.641, Mixed Models Analysis; Odds Ratio (OR) = 1.25, 90% CI 2-sided [0.57 to 2.74]
Statistical Analysis 2: Comparison: Group 2 DOR + IM DMPA vs Group 4 DOR + IUD; Week 4; Test type: Other; p = 0.204, Mixed Models Analysis; Odds Ratio (OR) = 1.57, 90% CI 2-sided [0.87 to 2.80]
Statistical Analysis 3: Comparison: Group 2 DOR + IM DMPA vs Group 4 DOR + IUD; Week 8; Test type: Other; p = 0.415, Mixed Models Analysis; Odds Ratio (OR) = 1.29, 90% CI 2-sided [0.77 to 2.15]
Statistical Analysis 4: Comparison: Group 2 DOR + IM DMPA vs Group 4 DOR + IUD; Week 12; Test type: Other; p = 0.027, Mixed Models Analysis; Odds Ratio (OR) = 2.23, 90% CI 2-sided [1.23 to 4.06]
Statistical Analysis 5: Comparison: Group 1 DOR + ETG vs Group 4 DOR + IUD; Week 2; Test type: Other; p = 0.274, Mixed Models Analysis; Odds Ratio (OR) = 1.86, 90% CI 2-sided [0.73 to 4.73]
Statistical Analysis 6: Comparison: Group 1 DOR + ETG vs Group 4 DOR + IUD; Week 4; Test type: Other; p = 0.065, Mixed Models Analysis; Odds Ratio (OR) = 1.83, 90% CI 2-sided [1.07 to 3.13]
Statistical Analysis 7: Comparison: Group 1 DOR + ETG vs Group 4 DOR + IUD; Week 8; Test type: Other; p = 0.252, Mixed Models Analysis; Odds Ratio (OR) = 1.72, 90% CI 2-sided [0.79 to 3.75]
Statistical Analysis 8: Comparison: Group 1 DOR + ETG vs Group 4 DOR + IUD; Week 12; Test type: Other; p = 0.002, Mixed Models Analysis; Odds Ratio (OR) = 2.61, 90% CI 2-sided [1.57 to 4.33]
Statistical Analysis 9: Comparison: Group 1 DOR + ETG vs Group 4 DOR + IUD; Week 20; Test type: Other; p = 0.460, Mixed Models Analysis; Odds Ratio (OR) = 0.78, 90% CI 2-sided [0.46 to 1.34]
Statistical Analysis 10: Comparison: Group 1 DOR + ETG vs Group 4 DOR + IUD; Week 24; Test type: Other; p = 0.019, Mixed Models Analysis; Odds Ratio (OR) = 1.59, 90% CI 2-sided [1.15 to 2.20]
Statistical Analysis 11: Comparison: Group 3 DOR + SC MPA vs Group 4 DOR + IUD; Week 2; Test type: Other; p = 0.061, Mixed Models Analysis; Odds Ratio (OR) = 2.16, 90% CI 2-sided [1.10 to 4.27]
Statistical Analysis 12: Comparison: Group 3 DOR + SC MPA vs Group 4 DOR + IUD; Week 4; Test type: Other; p = 0.106, Mixed Models Analysis; Odds Ratio (OR) = 1.64, 90% CI 2-sided [0.99 to 2.71]
Statistical Analysis 13: Comparison: Group 3 DOR + SC MPA vs Group 4 DOR + IUD; Week 8; Test type: Other; p = 0.144, Mixed Models Analysis; Odds Ratio (OR) = 1.77, 90% CI 2-sided [0.93 to 3.36]
Statistical Analysis 14: Comparison: Group 3 DOR + SC MPA vs Group 4 DOR + IUD; Week 12; Test type: Other; p = 0.011, Mixed Models Analysis; Odds Ratio (OR) = 2.37, 90% CI 2-sided [1.36 to 4.16]

3. Secondary Outcome: Number of Participants With HIV Viral Suppression (i.e. ART Efficacy)
Description: DOR-containing ART efficacy via HIV viral load <40 copies/mL
Time Frame: at 12-24 weeks after contraceptive initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 DOR + ETG | Group 2 DOR + IM DMPA | Group 3 DOR + SC MPA | Group 4 DOR + IUD | Group 5 DTG + DMPA
Number analyzed (Participants) | 21 | 21 | 22 | 19 | 21
Participants | 18 | 18 | 18 | 16 | 18

ADVERSE EVENTS:
Time Frame: Adverse event data were collected per participant from study enrollment to study exit, the median number of days were 141 days (IQR is 131.8, 217) or approximately 4.7 months
Arm/Group | Group 1 DOR + ETG | Group 2 DOR + IM DMPA | Group 3 DOR + SC MPA | Group 4 DOR + IUD | Group 5 DTG + DMPA
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/22 | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 1/22 | 1/19 | 0/21
Other Adverse Events (participants affected / at risk) | 20/21 | 20/21 | 21/22 | 18/19 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 DOR + ETG (N=21) | Group 2 DOR + IM DMPA (N=21) | Group 3 DOR + SC MPA (N=22) | Group 4 DOR + IUD (N=19) | Group 5 DTG + DMPA (N=21)
Motor vehicle accident (Injury, poisoning and procedural complications) | NA | NA | 0 | 1 | NA
Transient ischaemic attack (Nervous system disorders) | NA | NA | 1 | 0 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 DOR + ETG (N=21) | Group 2 DOR + IM DMPA (N=21) | Group 3 DOR + SC MPA (N=22) | Group 4 DOR + IUD (N=19) | Group 5 DTG + DMPA (N=21)
Gynaecological, etc. (Reproductive system and breast disorders) | 8 | 9 | 11 | 11 | 8
Neurological, eyes, etc. (Nervous system disorders) | 11 | 9 | 11 | 6 | 7
Gastrointestinal, etc. (Gastrointestinal disorders) | 7 | 9 | 8 | 5 | 3
Skin, alopecia, etc. (Skin and subcutaneous tissue disorders) | 6 | 5 | 6 | 1 | 3
Respiratory, etc. (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 7 | 4 | 4
Musculoskeletal, etc. (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 5 | 3
Ear, nose and throat (Ear and labyrinth disorders) | 2 | 6 | 1 | 2 | 2
Systemic, oral, oropharygyeal, etc. (General disorders) | 4 | 2 | 2 | 2 | 0
Cardiovascular, etc. (Cardiac disorders) | 1 | 0 | 1 | 2 | 4
Dyslipidaemia, haematology, etc. (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 0
Urogenital, etc. (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Motor vehicle accident, etc. (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
First, that not all participants adhered to their ART optimally limits exposure-outcome relationship ascertainments. Second, our timings of blood collection for doravirine analyses were suboptimal, resembling "random" time sampling; assuming this sampling is non-differential between the groups, our estimates will be biased towards the null. Third, the doravirine + etonogestrel implant group for hormone concentrations' outcome is compared to a historical group from a similar study but in Kenya.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04669678/Prot_SAP_ICF_000.pdf